CLINICAL TRIAL: NCT07148141
Title: Fertility Preservation for Patients With Breast Cancer: Altered Response to Ovarian Stimulation and Loss of Cholesterol Homeostasis in Ovarian Follicles
Brief Title: Impact of Breast Cancer on Human Folliculogenesis
Acronym: FERTICAN
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_BRUGNON_FERTICAN
Record Dates: First submitted 2025-08-19; First posted 2025-08-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Female; Infertility, Female
Keywords: oncofertility; Breast cancer; Fertility preservation; Folliculogenesis; Cholesterol biosynthesis
MeSH Terms: conditions — Infertility, Female; Breast Neoplasms | interventions — Ovulation Induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer patients (BC): Breast cancer subgroups (Triple-negative breast cancer (TN), Hormone-dependent breast cancer (HR+), HER2-amplified breast cancer (HER2+))
  Interventions: Other: Ovarian stimulation
- Oocyte donors (OD): Healthy women
  Interventions: Other: Ovarian stimulation

INTERVENTIONS:
Other: Ovarian stimulation — Ovarian stimulation before oocytes retrieval

SUMMARY:
Advances in cancer diagnosis and treatments have improved the 5-year survival rate for patients over the last decade. Nevertheless, cancer treatments frequently alter patient's fertility, thus compromising their ability to conceive a child after remission. Consequently, it is recommended to propose fertility preservation to patients before cancer therapy. The reference technique for preserving women's fertility the vitrification of mature oocytes after hormonal stimulation. In the context of cancer, different studies have shown that ovarian response to stimulation seems to be altered compared to healthy context, with a reduced number of mature oocytes collected, and altered oocyte quality, thus reducing the number of oocytes capable of producing a viable embryo. Hence, cancer seems to exert a deleterious impact on women's fertility. Nevertheless, the mechanisms by which the cancer may impair the ovarian functions are poorly understood. This innovative project aims to study the impact of breast cancer itself (the most frequent cancer in reproductive-aged women) on ovarian functions, and more precisely on the cholesterol biosynthesis pathway. Indeed, cholesterol homeostasis is essential for oocyte maturation and fertilization. The objectives of this study are i) to evaluate the impact of breast cancer on ovarian reserve and response to hormonal stimulation according to the molecular subtypes of breast cancer and ii) to evaluate the impact of breast cancer on ovarian cholesterol homeostasis in granulosa cells and follicular fluids.

This original approach will improve the understanding of the mechanisms underlying the impact of breast cancer on ovarian functions, and will have a strong clinical impact by helping to optimize fertility preservation strategies based on tumour molecular subtypes.

DETAILED DESCRIPTION:
Breast cancer patients (stratified into three molecular subgroups based on tumour hormonal status: HR+, HER2+, or triple-negative (TN)) and healthy oocyte donors (OD) are included in this study. During oocyte retrieval (for fertility preservation or oocyte donation), cumulus-oocyte complexes (COCs) are collected following ovarian stimulation. COCs are treated with hyaluronidase to separate the oocytes from surrounding cumulus granulosa cells. Clinical data regarding ovarian reserve and response to stimulation are collected.

Comparative analyses are conducted between breast cancer patients and oocyte donors, as well as between each molecular subgroup (TN vs. OD, HR+ vs. OD, HER2+ vs. OD). Following retrieval, granulosa cells and follicular fluids are collected. Total RNA is extracted from cumulus cells for RT-qPCR quantification of key enzymes and regulators involved in the cholesterol biosynthesis pathway. In parallel, cholesterol levels in follicular fluid are quantified using GC-MS/MS or FID-MS/MS.

This extended protocol enables both clinical and molecular comparisons to assess how breast cancer subtypes may differentially impact ovarian response and follicular environment

ELIGIBILITY:
Inclusion Criteria:

* Women above 18 years old and below 38 years old
* First hormonal stimulation cycle
* No dysovulation
* No cancer treatments prior fertility preservation (tumour resection, chemotherapy, radiotherapy)
* Women capable of giving written informed consent to participate in the research study
* Affiliated to social welfare service

Exclusion Criteria:

* Women below 18 years old and above 38 years old
* Endocrine disease
* Endometriosis
* Any cancer treatments prior fertility preservation (tumour resection, chemotherapy, radiotherapy)
* Previous hormonal stimulation cycle of less than six months

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Breast cancer patients and oocytes donors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Fertility preservation for patients with breast cancer: Altered response to ovarian stimulation and loss of cholesterol homeostasis in ovarian follicles | 65 months
  After oocyte retrieval, total RNA of granulosa cells from breast cancer patients and oocyte donors, will be extracted. Following retro transcription, qPCR will be performed

SECONDARY OUTCOMES:
Assessment of Anti-Mullerian Hormone levels | 36 months
  Ovarian reserve, assessed by Anti-Müllerian Hormone (AMH) levels, will be compared between oocyte donors and breast cancer patients according to molecular subtypes (TN, HR+, HER2+), BRCA mutation status, tumor grade, and lymph node involvement.
Assessment of antral follicle count | 36 months
  Ovarian reserve, assessed by antral follicle count, will be compared between oocyte donors and breast cancer patients according to molecular subtypes (TN, HR+, HER2+), BRCA mutation status, tumor grade, and lymph node involvement.
Total dose of FSH administered | 36 months
  Ovarian response parameters, assessed by the total dose of FSH administered, will be compared between oocyte donors and breast cancer patients according to molecular subtypes (TN, HR+, HER2+), BRCA mutation status, tumor grade, and lymph node involvement.
Number of harvested oocytes | 36 months
  Ovarian response parameters, assessed by the numver of harvested oocytes, will be compared between oocyte donors and breast cancer patients according to molecular subtypes (TN, HR+, HER2+), BRCA mutation status, tumor grade, and lymph node involvement.
Oocyte maturity | 36 months
  Ovarian response parameters, assessed by the number of mature oocytes, will be compared between oocyte donors and breast cancer patients according to molecular subtypes (TN, HR+, HER2+), BRCA mutation status, tumor grade, and lymph node involvement.
Oocyte atresia | 36 months
  Ovarian response parameters, assessed by the number of atretic oocytes, will be compared between oocyte donors and breast cancer patients according to molecular subtypes (TN, HR+, HER2+), BRCA mutation status, tumor grade, and lymph node involvement.
Impact of breast cancer on enzymes and regulators of the cholesterol biosynthetic pathway | 36 months
  Gene expression levels of enzymes (HMGCoA Réductase, SQLE, LSS, CYP51, DHCR7, DHCR24) and regulators (SREBP2, SCAP, INSIG, LXRa, LXRb) of the cholesterol biosynthesis will be assessed in cumulus cells by RT-qPCR and compared between breast cancer patients according to the molecular subtypes (TN, HR+, HER2+) and oocyte donors.
Quantification of cholesterol and its intermediates in follicular fluids of Breast Cancer patients and Oocytes Donors | 36 months
  Quantification of cholesterol and its intermediates will be assessed in follicular fluids by GC-MS/MS or GC-MS/FID and compared between breast cancer patients according to the molecular subtypes (TN, HR+, HER2+) and oocyte donors.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Brugnon, MD, PhD, HDR, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne Rhones-Alpes, France